CLINICAL TRIAL: NCT04503655
Title: Etude Multicentrique Évaluant L'efficacité D'une Intervention Visant À Réduire La Durée De Séjour Après L'implantation D'une Bioprothèse Aortique Par Voie Transfémorale
Brief Title: Multicenter Study Evaluating the Efficacy of an Intervention Aimed At Reducing the Length of Stay After Transfemoral Transcatheter Aortic Valve Implantation
Acronym: FAST-TAVI II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020/0185/HP
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Aortic Valve Stenosis; Cardiovascular Diseases
Keywords: TAVI; Aortic valve stenosis; Lenght-of-stay; Medico-economy
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: In this study, there is a randomization of the participating centres in two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The randomized centres in this group will be follow a training dedicated on implementation of "organizational" and "therapeutic" measures (for prevention and management of complications) to reduce lenght-of-stay after TF TAVI.
  Interventions: Other: Training
- Control group (No Intervention): The randomized centres in this group will not change their practices.

INTERVENTIONS:
Other: Training — Training dedicated on implementation of "organizational" and "therapeutic" measures (for prevention and management of complications) to reduce lenght-of-stay after TF TAVI.
  Arms: Intervention group

SUMMARY:
Since the first implantation of a percutaneous aortic bioprosthesis (TAVI) in 2002 (Cribier et al. Circulation 2002), TAVI occupies an increasing place in the management of aortic stenosis (AR) . Initially reserved for inoperable patients at high surgical risk, TAVI is also recommended in patients at intermediate risk, especially when a femoral approach (TF) is possible (Baumgartner et al. Eur Heart J. 2017).

Currently, there is no recommendation regarding length of stay after TAVI and practices are extremely heterogeneous. Despite the growing experience of centers, better patient selection and a reduction in complications, the length of stay after TAVI remains very high in France.

Faced with the great disparity observed between the centers, efforts are necessary to educate the centers in order to further reduce the length of stay after TF-TAVI. The aim of the study is to evaluate the effectiveness of an intervention based on training teams to reduce the length of stay after TF-TAVI.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years of age;
2. Patient hospitalized for TF-TAVI
3. Patient affiliated or benefiting from a health insurance scheme
4. Patient having read and understood the information letter and having signed the consent form.

Exclusion Criteria:

1. Proven pregnant woman (positive urine pregnancy test) or breastfeeding or absence of effective contraception (as defined by the WHO) or postmenopausal woman without confirmation diagnosis obtained (amenorrhea not medically induced for at least 12 months before the initiation visit) ; 1
2. Person deprived of their liberty by an administrative or judicial decision or person placed under the protection of justice / guardianship or curatorship
3. History of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participating in the protocol or preventing him from giving his informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1842 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of a multi-component organizational intervention | Year 1
  Proportion of patients benefiting from TF-TAVI with a length of stay less than or equal to 3 days.

SECONDARY OUTCOMES:
To evaluate the safety of the intervention | Day 30
  This outcome will be evaluated using :
  * the average length of stay,
  * the 30-day rehospitalization rate and
  * the 30-day death rate.
To evaluate the budgetary impact of the intervention | Year 1
  This outcome will be assessed using:
  * the hospital costs from the point of view of the hospital and
  * the financial gains for health insurance that would be associated with the generalization of the intervention in France.
To evaluate the implementation of the intervention | Year 1
  This outcome will be evaluated using the rate of adherence of the centers to the procedures aiming to reduce the length of stay (questionnaires)
To identify the factors associated with the effectiveness and safety of the intervention | Year 1
  This outcome will be assessed using factors associated with lengths of stay less than or equal to 3 days.

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - Hôpital privé Saint Martin, Caen
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Henri Mondor (AP-HP), Créteil
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHU de Limoges, Limoges
  - Hôpital privé Jacques Cartier, Massy
  - Clinique du Millénaire, Montpellier
  - Hôpital Bichat, AP-HP, Paris
  - Hôpital Européen Georges Pompidou (AP-HP), Paris
  - CHU de Poitiers, Poitiers
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - Clinique Pasteur, Toulouse
  - Clinique Saint Gatien, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Durand E, Beziau-Gasnier D, Michel M, Iung B, Tchetche D, Bonnet G, Lhermusier T, Gilard M, Souteyrand G, Bouleti C, Ohlmann P, Lefevre T, Beygui F, Chassaing S, Chevreul K, Eltchaninoff H; FAST-TAVI II; STOP-AS investigators. Reducing length of stay after transfemoral transcatheter aortic valve implantation: the FAST-TAVI II trial. Eur Heart J. 2024 Mar 14;45(11):952-962. doi: 10.1093/eurheartj/ehae081. PMID 38437633